CLINICAL TRIAL: NCT00300638
Title: Affective and Conative Changes in Alcoholism
Brief Title: Alcoholism: Emotion and Thinking
Status: Terminated | Type: Observational
Why Stopped: The study was terminated prematurely because of restrictions imposed by COVID-19.
Sponsor: Boston University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: H-24686; R01AA007112 (NIH); K05AA000219 (NIH)
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Alcoholism
Keywords: Alcoholism; Emotion; Cognition; Brain scans
MeSH Terms: conditions — Alcoholism | interventions — Magnetic Resonance Spectroscopy; Interviews as Topic; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 1- MRI and interviews: In our research, we are trying to understand where in the brain these emotional behaviors take place, and whether or not the brain functions differently for alcoholic and nonalcoholic individuals. We present emotional words and pictures on a computer screen, and using Magnetic Resonance Imaging (MRI) scans, we observe how the brain works when people purposefully respond to the words and pictures. Interviews, cognitive tests, and emotional measurements will also be done. Additionally, we are comparing brain structure and activation patterns in men and women, because there may be gender differences in responses to emotional stimuli.
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Behavioral: Interviews, cognitive tests, and emotional measurements

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging (MRI) — We present emotional words and pictures on a computer screen, and using MRI scans, we observe how the brain works when people purposefully respond to the words and pictures. Additionally, we are comparing brain structure and activation patterns in men and women, because there may be gender differences in responses to emotional stimuli.
Behavioral: Interviews, cognitive tests, and emotional measurements — We present emotional words and pictures on a computer screen, and using MRI scans, we observe how the brain works when people purposefully respond to the words and pictures. Additionally, we are comparing brain structure and activation patterns in men and women, because there may be gender differences in responses to emotional stimuli.

SUMMARY:
The purpose of this study is to determine whether long-term chronic alcoholism is associated with changes in emotional functioning and brain structure and function.

DETAILED DESCRIPTION:
This research investigates brain structure and function in alcoholics compared to healthy nonalcoholic individuals. Alcoholics have shown impairments in cognitive processing of emotional signals. Some alcoholics are impaired in social skills, and many are unable to implement the strategies for interpersonal interactions that they recommend for themselves. For example, alcoholics have difficulty interpreting non-verbal emotional cues and recognizing facial expressions of emotion. When listening to sentences, alcoholics also have some difficulty judging emotional intonations and emotional content. In our research, we are trying to understand where in the brain these emotional behaviors take place, and whether or not the brain functions differently for alcoholic and nonalcoholic individuals. We present emotional words and pictures on a computer screen, and using MRI scans, we observe how the brain works when people purposefully respond to the words and pictures. Additionally, we are comparing brain structure and activation patterns in men and women, because there may be gender differences in responses to emotional stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Male and female right-handed people 25 years of age or older.
* Participants either will have a past Diagnostic and Statistical Manual version IV (DSM-IV) diagnosis of alcohol dependence, or no such history at all.
* Participants will have signed an informed consent.

Exclusion Criteria:

* Pregnant women.
* Shrapnel or other metal in body (dental fillings OK)

Ages: 25 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Alcoholics and demographically equivalent healthy controls who have participated in one or more of our prior studies are contacted by telephone to determine whether or not they would like to participate again. Potential participants who have not previously been enlisted in any of our studies are recruited through fliers placed in the Boston Veterans Affairs Healthcare System, BU School of Medicine, and after-care programs in the Boston area, and through ads in local newspapers and web sites. For "new" participants, subject selection procedures include an initial prescreening telephone interview to determine identifying information such as age, level of education, health history, and history of alcohol and drug use and if eligible are invited to the laboratory for further screening and neuropsychological evaluations.
Sampling Method: Non-Probability Sample
Enrollment: 599 (Actual)
Dates: Start 2001-08 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Alcoholism's effects on thinking, behavior and brain functioning | several visits over approximately one month

CONTACTS AND LOCATIONS:
Overall Officials: Marlene O. Berman, PhD, Principal Investigator — Boston University
Locations (1):
- VA Hospital and Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Oscar-Berman M, Marinkovic K. Alcoholism and the brain: an overview. Alcohol Res Health. 2003;27(2):125-33. PMID 15303622